CLINICAL TRIAL: NCT06137495
Title: Immunoblot and Chemiluminescence Assays Versus ImmunoCap: Evaluation of Allergen Specific IgE in Egyptian House Dust Mites Allergic Rhinitis Patients
Brief Title: Immunoblot, Chemiluminescence and ImmunoCap Allergen Specific IgE Evaluation of in Allergic Rhinitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Noha M Hammad, MD, Associate Professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6489-8-11-2020
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Diagnoses Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allergic Rhinitis Patients (Experimental): House dust mites (HDMs) IgE in sera of allergic rhinitis patients (AR) who were monosensitized to mixed HDMs, identified by SPT, is assayed using immunoblotting, chemiluminescence, and ImmunoCAP assays to compare between the accuracy of both immunoblotting and chemiluminescence assays, and ImmunoCAP as gold standard
  Interventions: Diagnostic Test: Sensitization to House dust mites

INTERVENTIONS:
Diagnostic Test: Sensitization to House dust mites — The SPT is performed at the time of diagnosis and after six-months follow-up period. Serum specific IgE is measured by immunoblotting, chemiluminescence, and ImmunoCAP assays
  Other Names: Allergen skin prick testing (SPT); Measurement of serum specific IgE

SUMMARY:
In the present study the investigators assay house dust mites (HDMs) IgE in sera of allergic rhinitis patients (AR) using immunoblotting, chemiluminescence, and ImmunoCAP assays to compare between the accuracy of both immunoblotting and chemiluminescence assays, and ImmunoCAP as gold standard.

DETAILED DESCRIPTION:
All allergic rhinitits patients who were monosensitized to mixed HDMs, identified by SPT, will be subjected to complete history taking and assessment of the inclusion and exclusion criteria, performance of skin prick test and measurement of total serum IgE, measurement of specific IgE by Chemiluminescence Immunoassa, immunoblot assay and ImmunoCAP™ Phadiatop™. The patients will be followed-up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient consent.
2. Patient with (18-40) years age known to be allergic rhinitis.
3. Patient with IgE mediated allergic rhinitis (positive total IgE).
4. Patient with positive skin prick testing and monosensitized to HDM

Exclusion Criteria:

1. Patient refusal
2. Patients taking oral corticosteroid.
3. Patients taking anti-IgE injections.
4. Patients taking intranasal corticosteroid.
5. Patient with non- IgE mediated allergic rhinitis.
6. Patients with chronic diseases.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction of serum specific IgE | 6 months from diagnosis to end of Follow-up period
  Improvement of symptoms and signs of allergy
Conversion of SPT to negative | 6 months from diagnosis to end of Follow-up period
  Improvement of symptoms and signs of allergy

CONTACTS AND LOCATIONS:
Overall Officials: Noha M Hammad, MD, Principal Investigator — Faculty of Medicine, Zagazig University
Locations (1):
- Zagazig University Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No